CLINICAL TRIAL: NCT05969379
Title: Genetic Predisposition, Inflammation, and Neurodegeneration Biomarkers in Patients With Neurological Adverse Events of Immune Checkpoint Inhibitors: Correlation With Clinical Phenotypes and Outcome
Brief Title: Investigational Biomarkers for Neurological Immune-related Adverse Events
Acronym: NFL-ICI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL23_0712
Record Dates: First submitted 2023-07-20; First posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Neurological Disease
Keywords: Biomarkers; autoimmunity; immunotherapy side-effects; immune checkpoint inhibitors; neuroimmunology
MeSH Terms: conditions — Nervous System Diseases; Autoimmune Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Serum, plasma EDTA, whole blood, CSF, PBMC
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with neurological immune-related adverse events (n-irAEs): Patients developing neurological syndromes related to administration of any immune checkpoint inhibitors, including central nervous system disorders and neuromuscular toxicties
  Interventions: Genetic: Analysis of biomarkers and their correlation with clinical characteristics and outcome

INTERVENTIONS:
Genetic: Analysis of biomarkers and their correlation with clinical characteristics and outcome — This is a non-interventional study involving clinical data, neuroimaging analysis, and biological samples. Demographics and clinical data are collected in the database of the French Reference Centre. Additional or missing data will be obtained by contacting the referral physicians. All the neuroimages available will be analysed by dedicated software. Samples are already stored in biobank repositories and collected as part of "good clinical practice" in the diagnostic process of patients with suspected autoimmune encephalitis, meaning that the standard diagnostic and therapeutic approaches will not be altered in the selected study population. Patients have already gave explicit written consent for biological specimens sampling and storage at the "Centre de Ressources Biologiques des Hospices Civils de Lyon" (CRB-HCL) (including tissue, cells or biological fluids). Additional samples for genetic testing will be collected upon explicit written consent.

SUMMARY:
Neurological immune-related adverse events (n-irAEs) are an emerging group of disorders of patients with cancer treated with immune checkpoint inhibitors, presenting with heterogeneous clinical manifestations and of uncertain outcome. Novel genetic, inflammatory, and neurogenerative biomarkers could be associated with distinct phenotypes and different outcomes. To test this hypothesis, the study will provide: a phenotypic characterization and outcome assessment of patients with n-irAEs; the analysis of biomarkers of genetic predisposition (HLA and other immunity-related genes), inflammation (serum and cerebrospinal fluid [CSF] cytokines and autoantibodies, peripheral blood and CSF lymphocytes and other immune cells, neuroimaging), neurodegeneration (serum and CSF neurofilaments, neuroimaging) and their correlation with clinical features and outcome.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of n-irAEs

Exclusion Criteria:

* Presence of an alternative diagnosis explaining the neurological syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at least 18 years-old with a diagnosis of n-irAE
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Analysis of neurofilaments | At enrollment
  Neurofilaments will be analysed by MSD.
  Meso Scale Discovery Electrochemiluminescence (MSD) uses sandwich enzyme-linked immunosorbent assay (ELISA) method coupled with electro¬chemiluminescence (ECL) detection and plate array technology to provide highly sensitive and multiplexed detection of the analytes of interest (like neurofilaments) in a complex biological matrix.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de référence des syndromes neurologiques paranéoplasiques et encéphalites auto-immunes, Hôpital neurologique Pierre Wertheimer, Bron, France